CLINICAL TRIAL: NCT04187170
Title: Longitudinal Analysis of Right Ventricular Remodeling in Response to Prolonged Strength Training Using 3D-echocardiography
Acronym: FORCE-VD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Principal Investigator, Amir HODZIC, Principal investigator, University Hospital, Caen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-092
Record Dates: First submitted 2019-11-17; First posted 2019-12-05 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Cardiac Remodeling, Ventricular; Right Ventricular Hypertrophy
Keywords: Right ventricle; cardiac physiology; strength training; echocardiography
MeSH Terms: conditions — Ventricular Remodeling; Hypertrophy, Right Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy sedentary subjects exposed to the training program (Experimental)
  Interventions: Other: Strength physical training

INTERVENTIONS:
Other: Strength physical training — progressive high-load strength training over 6 months, consisting in repeated physical exercises to increase the muscular mass and force by altering concentric and eccentric muscle contractions against high resistance.

SUMMARY:
Right ventricular (RV) physiological remodeling in response to prolonged strength exercise remains poorly studied. This prospective, non-randomized, single-center study, proposes to follow 24 healthy sedentary volunteers who will benefit from a high-intensity pure resistance training program over a 6-month period. The volunteers, aged between 18 and 40 years old and male, will be recruited and evaluated at the University Hospital center of Caen Normandy. Cardiac remodeling in response to physical exercise will be analyzed by trans-thoracic echocardiography repeated during the follow-up. The physical impact of the training program will be assessed by a treadmill exercise test predicting maximal oxygen consumption (VO2max) before and after completing the training, and an isokinetic muscular test repeated every 3 months. Participants rest/activity cycles will be monitor before and after 3 months of training. The aim of the study is to demonstrate the existence of a physiologic RV remodeling in response to pure high-load resistance chronic exercise. The results will help to improve the understanding of the physiological RV response expected in strength athletes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years
* Male gender
* Agree to participate in the study (signature of consent).
* Affiliated to an insurance scheme or beneficiary

Exclusion Criteria:

* Female gender
* Inability to express consent
* Moderate physical activity over than 150 minutes or intensive physical activity over than 75 minutes per week on a regular basis for more than 6 consecutive months, according to the World Health Organisation criteria.
* Participation in competitive sports of ≥ II and / or B according to Mitchell's classification in the last 3 years.
* Ischemic and non-ischemic heart diseases
* Family history of unexplained sudden death
* Personal or family history of elastic tissue disease (Marfan syndrome and related)
* Chronic diseases incompatible with physical exercise at high intensity
* Personal history of chemotherapy and / or radiotherapy
* ≥ 1 cardiovascular risk factors
* use of doping substances
* Body mass index > 30 kg/m²
* Inclusion in another biomedical research protocol (during the present study or within 6 months before inclusion).

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Assessment of right ventricular volumes change over 6 months of sustained high-strength physical training. | Before the training starts and up to 6 months of follow-up
  Analysis of variation in echocardiographic measurements of RV volumes before and after training

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Caen, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pamart N, Drigny J, Azambourg H, Remilly M, Lahjaily K, Rocamora A, Tournoux F, Saloux E, Reboursiere E, Gauthier A, Hodzic A. Association between muscle strength gains and biventricular cardiac remodeling in response to high-intensity resistance training in healthy untrained males: a longitudinal study. BMC Sports Sci Med Rehabil. 2025 May 7;17(1):116. doi: 10.1186/s13102-025-01165-8. PMID 40336139
- [Derived] Pamart N, Drigny J, Azambourg H, Remilly M, Macquart M, Lefevre A, Lahjaily K, Parienti JJ, Rocamora A, Guermont H, Desvergee A, Ollitrault P, Tournoux F, Saloux E, Normand H, Reboursiere E, Gauthier A, Hodzic A. Effects of a 20-Week High-Intensity Strength Training Program on Muscle Strength Gain and Cardiac Adaptation in Untrained Men: Preliminary Results of a Prospective Longitudinal Study. JMIR Form Res. 2023 Oct 24;7:e47876. doi: 10.2196/47876. PMID 37874630
- See also: Abstract Journées Européennes de la Société Française de Cardiologie 2024 — https://doi.org/10.1016/j.acvd.2023.10.210
- See also: Effects of a 20-Week High-Intensity Strength Training Program on Muscle Strength Gain and Cardiac Adaptation in Untrained Men: Preliminary Results of a Prospective Longitudinal Study — http://pubmed.ncbi.nlm.nih.gov/37874630/